CLINICAL TRIAL: NCT05635799
Title: Virtual Reality Applied to the Evaluation and Rehabilitation of Locomotion - Study of Tolerance in the Lower Limb Amputee
Acronym: REVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CASILLAS CRBFC-E 2019
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Unilateral Amputation of the Lower Limb
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with lower limb amputations (Experimental)
  Interventions: Other: Analysis of walking on flat ground; Other: Hospital Anxiety Disorder Questionnaire; Other: Analysis of walking on slopes; Other: Group interview with a sociologist
- Healthy volunteers (Active Comparator)
  Interventions: Other: Analysis of walking on flat ground; Other: Hospital Anxiety Disorder Questionnaire; Other: Analysis of walking on slopes

INTERVENTIONS:
Other: Analysis of walking on flat ground — Analysis of walking on flat ground under different environmental conditions (visit 1)
Other: Hospital Anxiety Disorder Questionnaire — performed during the inclusion visit
Other: Analysis of walking on slopes — All assessments will be identical to the flat walking analysis: flat walking will be replaced by slope walking for all environmental conditions
Other: Group interview with a sociologist — Virtual reality feedback, accompanied by a confrontation of the patients' subjective experiences (group of 5 to 10 people)
  Arms: Subjects with lower limb amputations

SUMMARY:
The adaptability of the locomotor activity allows to face all the modifications of the immediate environment met in the daily activities. These situations become complex to apprehend for a person with a locomotor disability such as patients fitted with a lower limb amputation device. Thus, these adaptation capacities are essential to take into account in the rehabilitation process to maximize autonomy and reduce the risk of falls. For this purpose, the Quantitative Gait Analysis (QGA) allows to measure the impact of these constraining situations on the organization of gait patterns. However, this evaluation could be considerably optimized in current practice with the contribution of Virtual Reality (VR), by its immersive power which brings it closer to real life conditions (walking in a straight line, going up/down steps, taking into account visual and sound constraints, etc.). Eventually, this immersive approach by various VR environments could allow to improve the rehabilitation protocols in a personalized and secure way.

In this context, this project proposes to measure the tolerance of volunteers in a specific virtual environment and to quantify the modifications induced by this immersive environment, during a simple locomotor act (walking on flat ground) and complex (walking on a slope) in healthy volunteers, in order to evaluate the impact of VR on locomotion in a healthy population, and then in a second time in lower limb amputee patients

This monocentric study will take place on the Technological Investigation Platform of the Dijon Bourgogne University Hospital.

25 healthy volunteers and 25 lower limb amputees (transtibial or transfemoral) will be included in this study.

The participants will make 3 visits:

* Visit 1 (inclusion visit and analysis of walking on flat ground)
* visit 2 (analysis of walking on slopes): between 15 days and 1 month after visit 1
* visit 3 (group interview with a sociologist): only for patients within 45 days after visit 2

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Person who has given oral consent
* Male or female over the age of majority, < 80 years
* Person able to understand simple commands, conditioning instructions

Amputee patients:

* Person who has given oral consent
* Male or female over the age of majority, < 80 years
* Patients with unilateral transfemoral or transtibial amputation of the lower limb of any origin (traumatic, vascular, congenital or neoplastic) with a definitive device.
* Patients with stable locomotion with aids, without technical aids
* Person able to understand simple orders, conditioning instructions

Exclusion Criteria:

Healthy Volunteers:

* Person who is not affiliated or not a beneficiary of a social security system
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant, parturient or breastfeeding woman
* Major incapable or unable to express his consent
* Minor
* Person with locomotor disorders (orthopedic, neurological, vascular, cardiac...) and/or balance disorders that may significantly alter walking
* Person with a contraindication to wearing a virtual reality helmet (uncontrolled epilepsy, wound of an area that the helmet would cover, severe ophthalmological disorders etc.)

Amputee patients:

* Person who is not affiliated or not a beneficiary of a social security plan
* Person under legal protection (guardianship, trusteeship)
* Person subject to a legal protection measure
* Pregnant, parturient or breastfeeding woman
* Major incapable or unable to express his consent
* Minor
* Person with locomotor disorders (orthopedic, neurological, vascular, cardiac...) other than amputation that may significantly alter walking
* Persons with contraindications to wearing a virtual reality helmet (uncontrolled epilepsy, wounds in an area that the helmet would cover, severe ophthalmological disorders, etc.)
* Patients unable to participate in a group interview (qualitative study only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Percentage of healthy volunteers who completed the virtual reality experiment (flat walk) without complications | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France